CLINICAL TRIAL: NCT06676397
Title: Characterization of the Homeostatic Functions of Eosinophils in Asthma: An Exploratory Study
Brief Title: Homeostatic Roles of Eosinophils in Asthma
Acronym: HOMEOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024/877
Record Dates: First submitted 2024-10-11; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Asthma; Eosinophilic
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Severe Asthma Patients : Biologic Naïves (Other): Severe Asthma Patients : Biologic Naïves
  Interventions: Procedure: Blood Punction
- Severe Asthma Patients: Responders to Biologics (Other): Severe Asthma Patients: Responders to Biologics
  Interventions: Procedure: Blood Punction
- Severe Asthma Patients: Non Responders to Biologics (Other): Severe Asthma Patients: Non Responders to Biologics
  Interventions: Procedure: Blood Punction
- Mild asthmatics (Other): Mild asthmatics
  Interventions: Procedure: Blood Punction
- Healthy Controls (Other): Healthy Controls
  Interventions: Procedure: Blood Punction

INTERVENTIONS:
Procedure: Blood Punction — venous blood sampling

SUMMARY:
The HOMEOS study is an exploratory, observational, and monocentric research. It focuses on characterizing the homeostatic roles of eosinophils in severe asthma. The primary objective is to identify eosinophil subpopulations among different groups of severe asthmatic patients using flow cytometry. The study aims to advance understanding of eosinophil diversity, which could guide new therapeutic approaches .

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mild asthma with severe asthma (Biologic-naïve, responders to anti-eosinophil biologic therapies and resistant to anti-eosinophil biologic therapies), control subjects without asthma
* Signature of informed consent
* Affiliation with the French social security system

Exclusion Criteria:

* Non-eosinophilic asthma
* Coexistence of a chronic eosinophilic inflammatory condition other than asthma
* Other respiratory conditions (cystic fibrosis, COPD, allergic bronchopulmonary aspergillosis, etc.)
* Treatment with corticosteroids within 10 days prior to inclusion
* Active smoking or a smoking history of more than 20 pack-years
* Pregnant women
* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate with the study and/or with anticipated low cooperation as assessed by the investigator
* Subject without health insurance
* Subject currently in an exclusion period of another study or as indicated by the "national registry of volunteers."

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-04 (Estimated); Primary Completion 2026-12-04 (Estimated); Study Completion 2027-02-04 (Estimated)

PRIMARY OUTCOMES:
Flow cytometry based eosinophil phenotyping : Expression levels of cell markers CD62L, CD123, CD101, CD11b, CD193, CD125, Siglec-8 on blood eosinophils quantified by flow cytometry and expressed in % and MFI (mean fluorescence intensity) | at inclusion
  Expression levels of cell markers CD62L, CD123, CD101, CD11b, CD193, CD125, Siglec-8 on blood eosinophils quantified by flow cytometry and expressed in % and MFI (mean fluorescence intensity)